CLINICAL TRIAL: NCT00256737
Title: Omeprazole Versus Anti-reflux Surgery in the Long-term Management of Peptic Esophagitis - a 10 Year Follow up Study of Patients Previously Studied for 5 Years - A Nordic Multicentre Study
Brief Title: Sopran - Omeprazole Treatment Versus Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D9584C00004; SH OMG 0004
Record Dates: First submitted 2005-11-20; First posted 2005-11-22 (Estimated); Last update posted 2011-01-24 (Estimated); Status verified 2011-01

CONDITIONS: GERD
Keywords: Maintenance of healed erosive esophagitis
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — Omeprazole

INTERVENTIONS:
Drug: Omeprazole

SUMMARY:
The purpose of this study is to study gastritis, GI symptoms during long term omeprazole treatment

ELIGIBILITY:
Inclusion Criteria:

* Previous inclusion into Astra study I-635 and willing to continue for another 10 years,

Exclusion Criteria:

* Pregnancy or lactation; Woman planning pregnancy within 5 years; Suspected or confirmed malignancy; Documented eradication of Helicobacter pylori.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 219
Dates: Start 1998-01; Primary Completion 2005-10 (Actual); Study Completion 2005-10 (Actual)

PRIMARY OUTCOMES:
Determine the safety of omeprazole during long term treatment

SECONDARY OUTCOMES:
To investigate the long term control of reflux symptoms, healing of esophagitis and persistence of post fundoplication symptoms during long term treatment of omeprazole

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca GI Medical Science Director, MD, Study Director — AstraZeneca
Locations (13):
- Denmark (6):
  - Research Site, Aalborg
  - Research Site, Glostrup Municipality
  - Research Site, Hillerød
  - Research Site, Kolding
  - Research Site, Odense
  - Research Site, Roskilde
- Research Site, Kuopio, Finland
- Norway (3):
  - Research Site, Bergen
  - Research Site, Oslo
  - Research Site, Trondheim
- Sweden (3):
  - Research Site, Gothenburg
  - Research Site, Örebro
  - Research Site, Stockholm

REFERENCES:
- [Derived] Attwood SE, Ell C, Galmiche JP, Fiocca R, Hatlebakk JG, Hasselgren B, Langstrom G, Jahreskog M, Eklund S, Lind T, Lundell L. Long-term safety of proton pump inhibitor therapy assessed under controlled, randomised clinical trial conditions: data from the SOPRAN and LOTUS studies. Aliment Pharmacol Ther. 2015 Jun;41(11):1162-74. doi: 10.1111/apt.13194. Epub 2015 Apr 10. PMID 25858519